CLINICAL TRIAL: NCT05294835
Title: Impact of Ketamine on Epigenetic Age (IKEA)
Brief Title: Ketamine and Epigenetic Aging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Wild Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD-WH-001
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Depression; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: prospective, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine Infusion (Experimental): subanesthetic ketamine infusion (0.5mg/kg) over 2-3 weeks
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine infusion

SUMMARY:
This is a prospective, clinical pilot study (n=20) to evaluate the impact of a ketamine treatment for Major Depressive Disorder (MDD) or Post Traumatic Stress Disorder (PTSD) on epigenetic aging by the TruAge epigenetic age laboratory test.

DETAILED DESCRIPTION:
Subjects with MDD or PTSD will have a series of six ketamine infusions over two to three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-64 years old of any sex, gender orientation, and ethnicity
* Read, understand, and provide written informed consent in English,
* Meet criteria for a primary psychiatric diagnosis of Major Depressive Disorder (MDD) or Post-traumatic Stress Disorder (PTSD) for greater than 4 weeks,
* Have a history of at least 1 failed medication trial targeting MDD or PTSD
* Have a reliable form of transportation to lodging or home following the completion of each ketamine infusion treatment day,
* Be generally healthy, as assessed by medical history, physical examination (including vital signs), and clinical laboratory evaluations,
* Be of non-childbearing potential or utilizing an acceptable form of birth control (females-only)
* Report a pre-treatment symptom level of ≧15 on the PHQ-9 or ≧ 33 on the PCL-5
* Consent to participation in venipuncture, drug test, pregnancy test (for females) psychiatric evaluation, rating scale completion and ketamine infusion treatment series of six over the course of two to three weeks.

Exclusion Criteria:

* Delirium or dementia diagnosis,
* Unstable medical illness or clinically significant laboratory results,
* History of clinically significant cardiovascular disease or electrocardiogram (EKG) findings, or medical conditions that put the patient at high risk for possible cardiac side effects, or uncontrolled hypertension
* History of multiple adverse drug reactions,
* Current or past history of psychotic disorder or psychotic symptoms,
* Current manic symptoms,
* Active substance use disorders with the exception of nicotine and caffeine, within the past six months or any past history of ketamine or PCP abuse,
* Requirement of excluded medications that interact with ketamine,
* Pregnancy, breastfeeding or unacceptable means of birth control in a female of child-bearing age,
* Current acute suicidal or homicidal risk,
* Previous exposure to ketamine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age | Biological age will be compared from baseline to study completion, an average of five weeks
  DNA Methylation-derived epigenetic age

SECONDARY OUTCOMES:
Severity of Illness and baseline epigenetic age | Assessment will evaluate the correlation of data collected at baseline with data from after treatment is completed, on average five weeks
  Assess if severity of illness prior to treatment is associated with biological age before treatment
Severity of Illness and post-treatment epigenetic age | Assessment will evaluate the correlation of data collected at baseline with biological age assessed after treatment is complete, on average five weeks
  Assess if severity of illness, as measured by PHQ-9 (Patient Health Questionnaire-9) or PCL-5 (PTSD Checklist for DSM 5) prior to treatment is associated with biological age after treatment
Degree of Treatment Response | Assessment will compare the difference in PHQ-9/PCL-5 scores from baseline to after treatment with change in biological age from baseline to post-treartment.
  Assess if degree of treatment response to ketamine infusion, as measured by PHQ-9 (Patient Health Questionnaire-9) or PCL-5 (PTSD Checklist for DSM 5), is associated with change in biological age

CONTACTS AND LOCATIONS:
Locations (1):
- Wild Health, Lexington, Kentucky, United States

REFERENCES:
- [Background] Han LKM, Aghajani M, Clark SL, Chan RF, Hattab MW, Shabalin AA, Zhao M, Kumar G, Xie LY, Jansen R, Milaneschi Y, Dean B, Aberg KA, van den Oord EJCG, Penninx BWJH. Epigenetic Aging in Major Depressive Disorder. Am J Psychiatry. 2018 Aug 1;175(8):774-782. doi: 10.1176/appi.ajp.2018.17060595. Epub 2018 Apr 16. PMID 29656664
- [Background] Marcantoni WS, Akoumba BS, Wassef M, Mayrand J, Lai H, Richard-Devantoy S, Beauchamp S. A systematic review and meta-analysis of the efficacy of intravenous ketamine infusion for treatment resistant depression: January 2009 - January 2019. J Affect Disord. 2020 Dec 1;277:831-841. doi: 10.1016/j.jad.2020.09.007. Epub 2020 Sep 7. PMID 33065824
- [Derived] Dawson KL, Carangan AMJM, Klunder J, Carreras-Gallo N, Sehgal R, Megilligan S, Askins BC, Perkins N, Mendez TL, Smith RM, Dawson MS, Mallin MP, Higgins-Chen AT, Dwaraka VB. Epigenetic aging and DNA methylation biomarker changes following ketamine treatment in patients with MDD and PTSD: a pilot study. Transl Psychiatry. 2025 Oct 31;15(1):452. doi: 10.1038/s41398-025-03683-y. PMID 41173838
- See also: "GrimAge," an epigenetic predictor of mortality, is accelerated in major depressive disorder — https://www.nature.com/articles/s41398-021-01302-0